CLINICAL TRIAL: NCT00833456
Title: Non-interventional Clinical Study to Observe Improvement in Global Assessment of Functioning in Patients With Schizophrenia, Treated With Atypical Antipsychotics
Brief Title: NIS to Observe Improvement in Global Assessment of Functioning in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NSI-SER-2008/1
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Seroquel SR; atypical antipsychotics; assessment of functioning; GAF scale
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Seroquel SR: Patients whose symptoms are controlled with Seroquel SR and started with the therapy up to 1 month before the inclusion
- 2: Atypical antipsychotics: Patients whose symptoms are controlled with atypical antipsychotic in once daily formulation (excluding Seroquel SR) and started with the therapy up to 1 month before the inclusion

SUMMARY:
The purpose of the study is to monitor the general functional changes among patients with schizophrenia, treated with atypical antipsychotics dosed once daily for a period of 6 months.The primary study objective is to compare general functioning of patients with schizophrenia treated with Seroquel SR between baseline and the last study visit. The secondary study objectives are to compare general functioning of patients with schizophrenia treated with other atypical antipsychotic medicinal products administered once daily between baseline and the last study visit, monitoring of other indicators of clinical improvement, evaluation of patient compliance and assessment of occurrence of adverse effects

ELIGIBILITY:
Inclusion Criteria:

* patients have a diagnosis of schizophrenia, as defined by DSM-IV-TR
* patients' symptoms are controlled with Seroquel SR started up to 1 month before the inclusion
* or patients' symptoms are controlled with other atypical antipsychotic in once daily formulation started up to 1 month before the inclusion

Exclusion Criteria:

* patients who are treated with Seroquel SR or other antipsychotic more than 1 month
* patients with prescribed antipsychotic combinations
* pregnant women or women who are breast-feeding
* patients who have been treated with antipsychotics in depot formulations for the last two months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients visiting psychiatrist's practice
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To compare improvement in global assessment of functioning (using the GAF scale) between the baseline and the final study visit in the Seroquel SR-treated group. | three times: 0, 12 and 24 weeks after inclusion

SECONDARY OUTCOMES:
To assess improvement in global assessment of functioning (using the GAF scale) between the baseline and the final study visit in the group of patients treated with other atypical antipsychotics | three times: 0, 12 and 24 weeks after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pregelj, MD, PhD, Principal Investigator — Psihiatricna klinika Ljubljana, Studenec 48, 1260 Ljubljana
Locations (14):
- Slovenia (14):
  - Research Site, Begunje na Gorenjskem
  - Research Site, Brezovica pri Ljubljani
  - Research Site, Brežice
  - Research Site, Idrija
  - Research Site, Koper
  - Research Site, Ljubljana
  - Research Site, Maribor
  - Research Site, Nova Gorica
  - Research Site, Novo Mesto
  - Research Site, Ormož
  - Research Site, Postojna
  - Research Site, Radenci
  - Research Site, Sežana
  - Research Site, Vojnik